CLINICAL TRIAL: NCT02784223
Title: Diagnostic Value of 18F-Choline PET/CT in Patients With a Thyroid Nodule With an Indeterminate Cytology: Pilot Study
Acronym: CHOCOLATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Canceropôle Nord Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHOCOLATE
Record Dates: First submitted 2016-05-24; First posted 2016-05-27 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Thyroid Gland
Keywords: F18-choline; Surgery; Indeterminate; Thyroid node
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PET-CT with F18-choline (Experimental): PET-CT with F18-choline examination will be performed before surgery
  Interventions: Device: Radiation : PET-CT with F18-choline examination

INTERVENTIONS:
Device: Radiation : PET-CT with F18-choline examination — PET-CT with F18-choline examination will be performed before surgery

SUMMARY:
The purpose of the study is to investigate the contribution of PET-CT with F18-choline in the diagnosis of thyroid nodule with indeterminate cytology in order to guide the best indication of surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient with thyroid nodule ≥15 mm with an indeterminate cytology according to the Bethesda Classification 2008 (vesicular lesion of undetermined significance (Bethesda 3); follicular neoplasm or Hürthle cells (Bethesda 4); lesion suspicious for malignancy (Bethesda 5)), and to be operated on
* Patient affiliated to a social security scheme
* Informed consent and signed

Exclusion Criteria:

* Thyroid nodules <15 mm
* Coalescing nodules preventing proper individualization of targeted nodule;
* Thyroid nodule with non-diagnostic cytology (Bethesda 1), benign cytology (Bethesda 2) or malignant cytology (Bethesda 6)
* Hot thyroid nodule on the thyroid scan
* Major subject to a measure of legal protection or unable to consent
* Pregnant women / nursing
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2016-05; Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Sensitivity | Up to 4 months
  Sensitivity of 18F-choline PET to detect the cases of thyroid cancer among patients with thyroid nodule with an indeterminate cytology.
Specificity | Up to 4 months
  Specificity of 18F-choline PET to detect the cases of thyroid cancer among patients with thyroid nodule with an indeterminate cytology.

SECONDARY OUTCOMES:
Predictive diagnostic capabilities | Up to 4 months
  Diagnostic capabilities of 18F-Choline PET in predicting thyroid cancer
Duration for acquisition | Up to 4 months
  Determination of the optimal duration for the PET acquisition.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre François Baclesse, Caen, France

REFERENCES:
- [Derived] Ciappuccini R, Licaj I, Lasne-Cardon A, Babin E, de Raucourt D, Blanchard D, Bastit V, Saguet-Rysanek V, Lequesne J, Peyronnet D, Grellard JM, Clarisse B, Bardet S. 18F-Fluorocholine Positron Emission Tomography/Computed Tomography is a Highly Sensitive but Poorly Specific Tool for Identifying Malignancy in Thyroid Nodules with Indeterminate Cytology: The Chocolate Study. Thyroid. 2021 May;31(5):800-809. doi: 10.1089/thy.2020.0555. Epub 2020 Dec 23. PMID 33183159